CLINICAL TRIAL: NCT01681888
Title: Clinical Trial of Surface EMG Biofeedback for Children With Cerebral Palsy and Associated Movement Disorders
Brief Title: Surface EMG Biofeedback for Children With Cerebral Palsy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI for this trial, which has been terminated, is no longer employed by USC. After repeated attempts of contact, we are unable to identify the PI's current employment. We would therefore request close out of this clinical trial record.
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Michelle Cullen, Research Compliance Manager, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Biofeedback2012
Record Dates: First submitted 2012-07-19; First posted 2012-09-10 (Estimated); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Cerebral Palsy; Dystonia; Hypertonia; Spasticity; Movement Disorders
MeSH Terms: conditions — Cerebral Palsy; Dystonia; Muscle Hypertonia; Muscle Spasticity; Movement Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surface EMG Biofeedback (Experimental)
  Interventions: Device: Sanger EMG Biofeedback Device

INTERVENTIONS:
Device: Sanger EMG Biofeedback Device

SUMMARY:
Movement disorders such as dystonia, hypertonia, and spasticity interfere with or prevent voluntary movement. Studies have suggested that using biofeedback to increase awareness of muscle activation can improve motor function in patients with motor deficits. The investigators hypothesize that the daily use of a surface electromyographic (SEMG) biofeedback device for one month will improve motor function in children and young adults with dystonia, hypertonia, and/or spasticity. The SEMG biofeedback device is worn over the muscle(s) the subject has difficulty in controlling and provides vibratory feedback about muscle activation. Groups of children and young adults (ages 3-21), with dystonia, hypertonia, and/or spasticity will be asked to wear a small (approx 1 square inch) sensory feedback device on their affected muscle(s) for 5 hours a day for one month. The device will vibrate and emit a blue light when the muscle is activated. At the start of the experiment, subjects will be tested on the Goal Attainment Scale (GAS), the Pediatric/Adolescent Outcomes Data Collections Instruments (PODCI), and the Barry Albright Dystonia Scale (BAD). For one month, subjects will practice goals without device. After a month, subject will be assessed again and be given device to practice goals for a month. After one month, the subjects will be tested on the outcome measures again and return device.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy, or associated movement disorders such as dystonia, spasticity, and/or hypertonia
* Able to wear device for given amount of time

Exclusion Criteria:

* Unable to wear device for at least 5 hours day for a month.

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Goal Attainment Scale | Two months
  The Goal Attainment Scale measures function in each of 5 areas that are individually chosen by the parents or adolescents at the initial visit. Parents and/or adolescents are encouraged to choose 2 basic movement goals and 3 goals related to function.

CONTACTS AND LOCATIONS:
Overall Officials: Terence Sanger, MD, PhD, Principal Investigator — University of Southern California
Locations (1):
- Children's Hospital of Los Angeles, Los Angeles, California, United States